CLINICAL TRIAL: NCT04957732
Title: The Effect of Wound Irrigation With Irrisept Delivery System on Abscess Healing in Patients Presenting to the Emergency Department
Brief Title: The Effect of Wound Irrigation With Irrisept on Abscess Healing (Irrisept UF Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research facility was restructured and no longer treated subjects in the study population.
Sponsor: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20101227
Record Dates: First submitted 2021-06-14; First posted 2021-07-12 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Abscess
Keywords: Wound Irrigation
MeSH Terms: conditions — Abscess

STUDY DESIGN:
Intervention Model Description: The randomization methodology was controlled by the site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (SoC) (Active Comparator): For subjects randomized to the control group, Standard of Care (SoC), which was normal saline, was used.
  Interventions: Device: Standard of Care (SoC)
- Irrisept (Active Comparator): For subjects randomized to the investigational group, Irrisept was used.
  Interventions: Device: Irrisept Delivery System

INTERVENTIONS:
Device: Standard of Care (SoC) — SoC consisted of irrigation with normal saline, using the same proprietary abscess irrigation tip as the Irrisept arm. SoC was used at the initial visit and at each subsequent 48-hour visit interval (up to 96 hours) until abscess healing.
  Arms: Standard of Care (SoC)
Device: Irrisept Delivery System — Irrisept is a manual, self-contained irrigation device capable of producing 7-8 psi of pressure for effective wound cleansing and irrigation. Irrisept contents include the Chlorhexidine Gluconate (CHG) solution, a 450 mL bottle, and Irriprobe applicator or an abscess irrigation tip. The bottle design allows users to control the pressure of the solution through manual bottle compression. The device had an option for use with an Irriprobe applicator or an abscess irrigation tip. Irrisept was used at the initial visit and at each subsequent 48-hour visit interval (up to 96 hours) until abscess healing.
  Other Names: Irrisept
  Arms: Irrisept

SUMMARY:
The purpose of this study was to evaluate the safety and effectiveness of Irrisept compared to standard of care treatment of skin and soft tissue infections in the form of abscesses.

DETAILED DESCRIPTION:
After being informed about the trial and potential risks, subjects completed an informed consent form prior to participation. After eligibility criteria was verified, an initial wound assessment examination was performed. Subjects were then randomized to the Irrisept or Standard of Care treatment group. At intervals of 48 hours (up to 96 hours) later, abscesses were assessed until healing occurred. If the subject required antibiotics, this was recorded, as well as results from the wound and Methicillin-resistant Staphylococcus Aureus (MRSA) cultures.

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompetent individuals, 12 years of age or older with an uncomplicated abscess

   1. Uncomplicated abscess is defined as ≤8 cm of induration (defined as firmness to touch) at the greatest diameter.
   2. ≤4 cm of surrounding erythema (surrounding redness).
2. Defined area of central fluctuance may or may not be present.
3. Patient must be able to answer questions.
4. Patient must be medically stable as defined by the emergency department physician.
5. Patient must participate voluntarily in the study.

Exclusion Criteria:

1. Currently receiving antibiotics or received antibiotics within the last 72 hours.
2. Evidence of systemic infection (fever, aches, chills, nausea).
3. Requires admission to the hospital for infection or for any other reason(s).
4. Abscess caused by a human or animal bite.
5. Prior history of hypersensitivity or allergy to Chlorhexidine Gluconate (CHG).
6. Immunodeficiency (examples: HIV positive, Crohn's disease, systemic lupus erythematosus, Addison's disease, psoriasis, splenectomy, leukemia, cancer (on chemotherapy)).
7. Currently on any immune-modifying medication (examples - prednisone, antivirals).
8. History of chronic skin infection (3 or more in the past year).
9. Chronic medical problem (for example, end-stage heart, liver, kidney or lung disease, diabetes mellitus, peripheral vascular disease, history of organ transplant).
10. Mental illness, including but not limited to, substance abuse, dementia, schizophrenia or mentally handicapped or challenged.
11. Incarcerated.
12. Patient is pregnant or thinks she may be pregnant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Petrik, MD, Principal Investigator — University of Florida/Shands Emergency Department
Locations (1):
- University of Florida, Shands Emergency Department, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2010 to November 2011, patients with skin and soft tissue infections, in the form of abscesses, were recruited from Shands Emergency Department at the University of Florida.
Pre-assignment Details: The planned sample size was 107 subjects enrolled in each arm. However, during the study, the site rearranged their ED and no longer treated abscesses. As a result, the study was terminated early after enrolling 35 subjects. Of those, 19 were on SoC and 16 were on Irrisept. A total of 30 subjects completed the study, with 12 subjects on Irrisept and 18 on SoC. For the 5 subjects that did not complete the study, 4 were on Irrisept and 1 on SoC.
Groups:
- Standard of Care (SoC): For subjects randomized to the control group, Standard of Care (SoC), which was normal saline, was used.
  SoC consisted of irrigation with normal saline, using the same proprietary abscess irrigation tip as the Irrisept arm. SoC was used at the initial visit and at each subsequent 48-hour visit interval until abscess healing.
- Irrisept: For subjects randomized to the investigational group, Irrisept was used.
  Irrisept contents include the Chlorhexidine Gluconate (CHG) solution, a 450 mL bottle, and Irriprobe applicator or an abscess irrigation tip. The device has an option for use with an Irriprobe applicator or an abscess irrigation tip. Irrisept was used at the initial visit and at each subsequent 48-hour visit interval until abscess healing.
Period: Overall Study
Arm/Group | Standard of Care (SoC) | Irrisept
Started | 19 | 16
Completed | 18 | 12
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Population: A total of 35 subjects were consented and randomized. There were no (0) screen failures. There were 16 subjects randomized to Irrisept and 19 to SoC. Of these, 12 subjects randomized to Irrisept and 18 subjects randomized to SoC completed the study.
Groups:
- Standard of Care (SoC): For subjects randomized to the control group, Standard of Care (SoC) (normal saline) was used at the initial visit and at each subsequent 48-hour visit interval (up to 96 hours) until abscess healing.
- Irrisept: For subjects randomized to the investigational group, Irrisept was used at the initial visit and at each subsequent 48-hour visit interval (up to 96 hours) until abscess healing.
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | Irrisept | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  Age - Known: <=18 years | 0 | 0 | 0
  Age - Known: Between 18 and 65 years | 18 | 12 | 30
  Age - Known: >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 8 | 7 | 15
  Female | 9 | 6 | 15
  Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Used Oral Antibiotics
Description: Oral antibiotic use was used to determine if the use of pressurized irrigation with Irrisept in uncomplicated abscesses improved wound healing when compared to pressurized irrigation with SoC (normal saline).
Time Frame: 24, 48, 72 & 96-hour visit intervals
Population: There were 4 timepoints for assessing abscess wound healing with the use of oral antibiotics: 24, 48, 72 & 96 hours.
Measure: Number; unit: participants
Groups:
- Standard of Care (SoC): For subjects randomized to SoC, normal saline was used.
  Assessments were made at the initial visit and at each subsequent 24-hour visit interval (up to 96 hours) until abscess healing.
- Irrisept: For subjects randomized to the investigational group, Irrisept was used.
  Assessments were made at the initial visit and at each subsequent 24-hour visit interval (up to 96 hours) until abscess healing.
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
participants
  Number of Subjects Requiring Oral Antibiotics at 24-hour Follow-up | 1 | 0
  Number of Subjects Requiring Oral Antibiotics at 48-hour Follow-up | 2 | 1
  Number of Subjects Requiring Oral Antibiotics at Follow-up : 72-hour Follow-up | 1 | 0
  Number of Subjects Requiring Oral Antibiotics at Follow-up : 96-hour Follow-up | 0 | 1

2. Primary Outcome: Abscess Wound Healing Determined By Wound Improvement Score
Description: Wound improvement assessments were used to determine if the use of pressurized irrigation with Irrisept in uncomplicated abscesses improved wound healing when compared to pressurized irrigation with SoC (normal saline). Wound improvement was assessed via a clinician's discretion, according to a 5-point Likert scale: 1 = clinically resolved, no signs of active infection; 2 = markedly improved, resolving infection and healing; 3 = improved with some remaining signs of active infection; 4 = unchanged, stable without signs of worsening clinical infection and; 5 = worsening conditions. The results are shown using a chi-squared test, as an average Likert score compared between the 2 arms.
Time Frame: Abscess wound healing, assessed by wound improvement, was reviewed at the 48-hour visit.
Population: 5 scale units were analyzed. These include: 1 = clinically resolved, no signs of active infection; 2 = markedly improved, resolving infection and healing; 3 = improved with some remaining signs of active infection; 4 = unchanged, stable without signs of worsening clinical infection and; 5 = worsening conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard of Care (SoC): For subjects randomized to SoC, normal saline was used.
  Assessments were made at the initial visit and 48-hour visit interval.
- Irrisept: For subjects randomized to the investigational group, Irrisept was used.
  Assessments were made at the initial visit and 48-hour visit interval.
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
score on a scale | 2.88 (0.93) | 2.50 (0.62)

3. Primary Outcome: Abscess Wound Healing Determined By Exudation Score
Description: Exudation assessments were used to determine if the use of pressurized irrigation with Irrisept in uncomplicated abscesses improved wound healing when compared to pressurized irrigation with SoC (normal saline). Exudation was assessed via a clinician's discretion, according to a 5-point Likert scale: 1 = none; 2 = scant; 3 = minimal; 4 = moderate and; 5 = copious. The results are shown using a chi-squared test to compare the means at baseline and 48-hours. A two-tailed t-test was conducted for the mean improvement.
Time Frame: Abscess wound healing, assessed by exudation, was reviewed at baseline and the 48-hour visit.
Population: 5 scale units were analyzed. These include: 1 = none; 2 = scant; 3 = minimal; 4 = moderate and; 5 = copious.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
score on a scale
  Baseline | 2.31 (1.21) | 2.40 (1.43)
  48-Hour Follow-up Visit | 2.00 (1.00) | 2.10 (1.44)

4. Primary Outcome: Abscess Wound Healing Determined By Pain Score
Description: Pain assessments were used to determine if the use of pressurized irrigation with Irrisept in uncomplicated abscesses improved wound healing when compared to pressurized irrigation with SoC (normal saline). Pain was assessed using a Visual Analogue Scale (VAS). The scale was measured in centimeters (cm) which ranged between 0 cm ("no pain" at the far left) to 9.5 cm ("most severe pain" at the far right). Subjects marked their pain rating on the scale with an "X". The distance from the beginning of the scale (far left) to the "X" was measured in cm. The mean VAS score was assessed at baseline and at the 48-hour follow-up visit. The overall mean improvement was compared between the 2 arms using two-tailed t-tests.
Time Frame: Abscess wound healing, assessed by pain, was reviewed at baseline and the 48-hour visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
units on a scale
  Baseline | 5.27 (2.79) | 6.33 (2.42)
  48-Hour Follow-up | 3.80 (3.08) | 3.91 (3.30)

5. Secondary Outcome: Oral Antibiotic Use Required, Determined By Erythema Area Size
Description: Erythema was assessed to determine if the use of Irrisept reduced or eliminated the need for oral antibiotics in uncomplicated abscesses. The mean circumference of the erythema area, measured in centimeters (cm), was assessed at baseline and 48-hours later. This was performed by the clinician drawing a circle with a marker around the area of redness surrounding the abscess. Mean improvement was compared between the 2 arms using two-tailed t-tests.
Time Frame: The need for oral antibiotics, assessed by erythema, was reviewed at baseline and the 48-hour visit.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
centimeters (cm)
  Baseline | 4.01 (2.44) | 3.25 (2.34)
  48-hour Follow-up | 3.41 (4.85) | 1.70 (1.27)

6. Secondary Outcome: Oral Antibiotic Use Required, Determined By Induration (Abscess Area Size)
Description: Induration or abscess size was assessed to determine if the use of Irrisept reduced or eliminated the need for oral antibiotics in uncomplicated abscesses. The need for oral antibiotics, assessed by the mean induration or abscess size (measured in cm), was reviewed at baseline and the 48-hour visit. Mean improvement was compared between the 2 arms using two-tailed t-tests.
Time Frame: 48-hours after baseline
Population: Induration was assessed at baseline and the 48-hour follow-up visit. The length and width (in centimeters) of the abscess was used to measure the wound area (induration). For each subject, the difference in area between the two timepoints was used to find the mean improvement for both arms.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
centimeters (cm)
  Baseline | 12.263 (10.03) | 10.238 (8.00)
  48-Hour Follow-up | 8.843 (8.53) | 5.875 (4.14)

7. Secondary Outcome: Oral Antibiotic Use Required Due To Warmth
Description: Warmth was assessed to determine if the use of Irrisept reduced or eliminated the need for oral antibiotics in uncomplicated abscesses. Clinicians recorded whether the abscess was warm for each subject initially and after 48 hours.
Time Frame: The need for oral antibiotics, assessed by warmth, was reviewed at baseline and the 48-hour visit.
Population: Warmth was assessed at baseline and the 48-hour follow-up visit. Chi-square tests for answers "yes" or "no" were run at the baseline and 48-hour follow-up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
Participants
  Baseline: Yes | 14 | 8
  Baseline: No | 4 | 4
  48-Hour Follow-up: Yes | 9 | 4
  48-Hour Follow-up: No | 9 | 8

8. Secondary Outcome: Oral Antibiotic Use Required Due To Fluctuance
Description: The presence of fluctuance was assessed to determine if the use of Irrisept reduced or eliminated the need for oral antibiotics in uncomplicated abscesses. Clinicians recorded whether fluctuance was present for each subject initially and after 48 hours.
Time Frame: The need for oral antibiotics, assessed by fluctuance, was reviewed at baseline and the 48-hour visit.
Population: Fluctuance was assessed at baseline and the 48-hour follow-up visit. Chi-square tests for answers "yes" or "no" were run at the baseline and 48-hour follow-up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
Participants
  Baseline: Yes | 8 | 5
  Baseline: No | 10 | 7
  48-hour Follow-up: Yes | 4 | 2
  48-hour Follow-up: No | 14 | 10

9. Other Pre Specified Outcome: Oral Antibiotic Use Required Due To Results of MRSA/Wound Culture
Description: The tertiary objective was to determine if the use of pressurized irrigation with Irrisept in uncomplicated abscesses improved wound healing in patients that have MRSA-positive wounds compared to pressurized irrigation with normal saline. No data was collected towards this objective; thus, the success or failure of this endpoint was not assessed.
  To be compliant with the CT.gov template, although the information is incorrect and no data was captured this outcome, data was entered for Irrisept subjects.
Time Frame: 0 days
Population: 0
Groups:
- Standard of Care: For subjects randomized to SoC, normal saline was used.
  Assessments were made at the initial visit and 48-hour visit interval.
Arm/Group | Standard of Care | Irrisept
Number analyzed (Participants) | 0 | 0

10. Post Hoc Outcome: Worsening Symptoms Causality
Description: Causality for each worsening event was determined by using the following categories: 'related', 'possibly related', 'unlikely related', 'unrelated' or 'unknown'.
Time Frame: Baseline and up to 48-hours later
Population: There was a total of 42 AEs for which causality assessments were made; 28 AEs were from subjects on SoC and 14 were from subjects on Irrisept.
Measure: Count of Units; unit: Total Number of Worsening Symptoms
Units Other Than Participants: Total Number of Worsening Symptoms
Groups:
- Standard of Care (SoC): For subjects randomized to SoC, normal saline was used.
  Assessments were made, beginning at the time of informed consent, until study completion.
- Irrisept: For subjects randomized to the investigational group, Irrisept was used.
  Assessments were made, beginning at the time of informed consent, until study completion.
Arm/Group | Standard of Care (SoC) | Irrisept
Number analyzed (Participants) | 18 | 12
Number analyzed (Total Number of Worsening Symptoms) | 28 | 14
Total Number of Worsening Symptoms
  Related Worsening Symptom | 0 | 0
  Possibly Related Worsening Symptom | 10 | 2
  Unlikely Related Worsening Symptom | 14 | 7
  Unrelated Worsening Symptom | 3 | 5
  Unknown Relation Worsening Symptom | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reviewed, beginning at baseline, up to study completion 48 hours later.
Description: The protocol did not outline procedures to capture AEs, as the primary purpose was to assess the primary and secondary endpoints. Therefore, AEs were assessed as a post-hoc analysis. Worsening of any symptoms from baseline were considered AEs. The categories of AEs included pain, vomiting, exudation, depth, erythema, swelling, induration, fluctuance, warmth, & signs of active infection. All cause mortality and serious adverse events were not collected nor assessed.
Groups:
- Standard of Care (SoC): For subjects randomized to SoC, normal saline was used.
  Assessments were made anytime after consent, while the study participated in the trial.
- Irrisept: For subjects randomized to the investigational group, Irrisept was used.
  Assessments were made anytime after consent, while the study participated in the trial.
Arm/Group | Standard of Care (SoC) | Irrisept
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 12/18 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=18) | Irrisept (N=12)
All Worsening Symptoms (Infections and infestations) | 12 (28) | 6 (14) — The categories of worsening symptoms include pain, vomiting, exudation, depth, erythema, swelling, induration, fluctuance, warmth, and signs of active infection.
Pain (Infections and infestations) | 4 (4) | 0 (0) — The worsening symptom was pain.
Vomiting (Infections and infestations) | 1 (1) | 0 (0) — The worsening symptom was vomiting.
Erythema (Infections and infestations) | 5 (5) | 1 (1) — The worsening symptom was erythema.
Swelling (Infections and infestations) | 2 (2) | 3 (3) — The worsening symptom is swelling.
Exudation (Infections and infestations) | 4 (4) | 2 (2) — The worsening symptom is exudation.
Depth (Infections and infestations) | 1 (1) | 4 (4) — The worsening symptom is depth.
Induration (Infections and infestations) | 6 (6) | 1 (1) — The worsening symptom is induration.
Fluctuance (Infections and infestations) | 1 (1) | 0 (0) — The worsening symptom is fluctuance.
Active Infection (Infections and infestations) | 1 (1) | 3 (3) — The worsening symptom is active infection.
Warmth (Infections and infestations) | 2 (2) | 0 (0) — The worsening symptom is warmth.
Redness (Infections and infestations) | 1 (1) | 0 (0) — The worsening symptom is redness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2012-07-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT04957732/Prot_001.pdf